CLINICAL TRIAL: NCT00188175
Title: A Phase II Study of Preoperative Intensity-Modulated Radiation Therapy For Lower Limb Soft Tissue Sarcoma
Brief Title: IMRT Lower Limb Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ontario Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UHN REB 03-0107-C
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMRT for lower limb soft tissue sarcoma (Experimental)
  Interventions: Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Radiation: Intensity Modulated Radiation Therapy — Pre-op Intensity Modulated Radiation Therapy for lower limb soft tissue sarcoma.

SUMMARY:
Intensity-modulated radiation therapy may make wound healing problems less likely by 1)precisely shaping the region of high radiation dose to the shape of the tissue which harbours tumour cells, and 2) precisely shaping the regions of low radiation dose to the shapes of the normal tissues which are more sensitive to radiation effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven soft tissue sarcoma
* Lesion lies between the iliac crest (hipbone) and the ankle
* Lesion is newly diagnosed
* Assessed by radiation oncologist and surgical oncologist

Exclusion Criteria:

* Benign histologies
* Histologies generally treated with chemotherapy
* Prior or recurrent cancer, except nonmelanomatous skin cancer or carcinoma in-situ of the cervix

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2003-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Major wound complications within 120 days following surgery | 120 days post-op

SECONDARY OUTCOMES:
Assess acute and late radiation toxicity including limb edema | up to120 days

CONTACTS AND LOCATIONS:
Overall Officials: Brian O'Sullivan, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada